CLINICAL TRIAL: NCT06453174
Title: CLinical Utility of Early Intervention Including the 5-Step Precision Medicine (5SPM) Method in First-episode Psychosis: The CLUMP Project
Acronym: CLUMP
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI23/00582
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Psychosis
Keywords: Psychotic Disorders; Personalised Precision Psychiatry; Pharmacogenetics; First-episode psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort one: A prospective sample of patients with a first episode psychosis referred over 18 months to the new early intervention in psychosis programme of Personalised Precision Psychiatry called PRINT - PRevention and early INTervention in mental health - at Salamanca University Healthcare Complex (CAUSA) in Salamanca, Spain.
  Interventions: Other: Adherence to the first prescribed antipsychotic medication
- Cohort two: A retrospective, consecutive (in reverse chronological order as registered in CAUSA electronic health records) sample of patients who suffered a first-episode psychosis before the implementation of PRINT.
  Interventions: Other: Adherence to the first prescribed antipsychotic medication
- Cohort three: For additional comparative purposes, we shall analyse environmental, clinical and pharmacogenetic information of patients with psychotic disorders of more than five years of evolution or with other mental disorders, whose data are currently stored, and ethically approved for research use, in our Unit of Pharmacogenetics and Precision Medicine at CAUSA.

INTERVENTIONS:
Other: Adherence to the first prescribed antipsychotic medication — We shall compare adherence to the first prescribed antipsychotic medication and pragmatic clinical and functional outcomes between two cohorts of patients with first-episode psychosis. One cohort will be comprised of patients treated before the implementation of an early intervention in psychosis model of Personalised Precision Psychiatry including pharmacogenetics, and the other of patients treated under this new model. Also, we shall compare the pharmacogenetic profiles and possible phenocopies (variations of phenotypes produced environmentally, e.g., due to polypharmacy, rather than genetically) between these first episode psychosis patients and a national cohort of patients with longer-term psychotic disorders or with other mental health conditions, to evaluate potential implications for clinical management at different stages of a psychotic illness, and across mental disorders.
  Groups: Cohort one; Cohort two

SUMMARY:
CLUMP is a project of translational research that intends to bridge the gap between what we already know about pharmacogenetics of antipsychotic drugs and what we still do to treat patients with first-episode psychosis (FEP). We aim to improve the adherence to antipsychotic drugs and, therefore, the outcomes of patients with FEP. To achieve this aim, our objectives are to: (1) Introduce a pioneering early intervention model of Personalised Precision Psychiatry, including pharmacogenetics, for patients with FEP; (2) ascertain whether such a model can reduce the elevated discontinuation rates of antipsychotic medications in this group; (3) assess the impact of this model on pragmatic efficacy and functional measures; (4) determine whether this innovation can bring cost benefit; and (5) establish a blueprint for implementing this precision model nationally and internationally. We shall compare all-cause discontinuation rates of the first prescribed antipsychotic medication (primary outcome), discontinuation rates by causes, pragmatic efficacy and tolerability measures, functional outcomes, and healthcare costs between two cohorts of patients with FEP followed for one year. One cohort will be comprised of patients treated before the implementation of the early intervention model of Personalised Precision Psychiatry, and the other of new patients treated under this model. Also, we shall compare pharmacogenetic information, and its implications for clinical management, between these patients and another national cohort of patients with either longer-term psychotic disorders or other mental health problems.

ELIGIBILITY:
Inclusion Criteria

* Patients with a diagnosis of first-episode psychosis, either non-affective or affective.
* Patients aged 12-35 years.
* Patients followed by clinical services for at least one year, or earlier if there was evidence of antipsychotic treatment discontinuation.
* For cohort one: Patients and/or their family or legal representatives must provide written consent to take part in the CLUMP Project, including pharmacogenetics analysis.
* For cohort two: This will not be a mandatory inclusion criterion, but all patients will be approached by our research team seeking their consent to obtain their pharmacogenetic profile for research purposes.

Exclusion Criteria

* Patients with first-episode psychosis due to organic causes, for example, brain diseases such as Huntington's and Parkinson's disease, HIV, syphilis, dementia, brain tumours or cysts, or brain injury.
* Patients with moderate to severe intellectual disability.
* Patients who plan to reside (cohort one) or spent (cohort two) most of the one-year follow-up period in a locality outside of the PRINT's catchment area.

Ages: 12 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Cohort one: A prospective sample of patients with a first episode psychosis referred over 18 months to the new early intervention in psychosis programme of Personalised Precision Psychiatry called PRINT - PRevention and early INTervention in mental health - at Salamanca University Healthcare Complex (CAUSA) in Salamanca, Spain.
  Cohort two: A retrospective, consecutive (in reverse chronological order as registered in CAUSA electronic health records) sample of patients who suffered a first-episode psychosis before the implementation of PRINT.
  Cohort three: For additional comparative purposes, we shall analyse environmental, clinical and pharmacogenetic information of patients with psychotic disorders of more than five years of evolution or with other mental disorders, whose data are currently stored, and ethically approved for research use, in our Unit of Pharmacogenetics and Precision Medicine at CAUSA.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause discontinuation | 30 months
  The CLUMP Project will gauge treatment adherence by tracking the cessation of initially prescribed antipsychotic medication, determined by either patients or treating clinicians. Discontinuation rates over a one-year follow-up period and the average time until discontinuation will be examined. For cohort one, follow-up begins when antipsychotic medication is prescribed based on pharmacogenetic guidance from the 5SPM method, while for cohort two, it starts at the time of the first antipsychotic prescription. Discontinuation is defined as the first day of a minimum 2-week interruption of the initially prescribed antipsychotic. Discontinuation dates will be extracted from clinical records, with approximations utilized if necessary.

SECONDARY OUTCOMES:
Pragmatic efficacy, tolerability, and functional outcome measures | 30 months
  In both cohorts, we'll gather data on practical effectiveness, tolerability, and functional outcomes. This encompasses monitoring hospital admissions, ER visits, and outpatient clinic attendance during follow-up, as well as changes in medications, antipsychotic dose adjustments (using chlorpromazine dose equivalents), side effects (including BMI impact), and resumption of work or academic activities. Cohort one patients will additionally complete the EQ-5D-5L questionnaire to assess overall improvement and guide treatment decisions at month 6. They'll also undergo assessments using various scales including PANSS, Calgary Depression Rating Scale, BNSS, and UKU side effects rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Pérez Sánchez-Toledo, PhD MD, Principal Investigator — Instituto de Investigación Biomédica de Salamanca
Locations (1):
- Instituto de Investigación Biomédica de Salamanca (IBSAL), Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided